CLINICAL TRIAL: NCT05311189
Title: Study of HLX10, Trastuzumab and Chemotherapy in First-line Treatment of HER2-positive Recurrent/Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, doctor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10GCIIT01
Record Dates: First submitted 2022-03-23; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: HER2-positive Gastric Cancer
MeSH Terms: interventions — Trastuzumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX10, Trastuzumab and Chemotherapy (Experimental): HLX10, Trastuzumab and Chemotherapy in First-line Treatment of HER2-positive Recurrent/Metastatic Gastric Cancer
  Interventions: Drug: HLX10, Trastuzumab and Chemotherapy

INTERVENTIONS:
Drug: HLX10, Trastuzumab and Chemotherapy — HLX10 4.5mg/kg, IV, q3weeks, Day 1 trastuzumab 6mg/kg (8mg loading dose), IV, q3weeks, Day 1 S1 40mg/m2, PO, BID, Day 1-14 oxaliplatin 100mg/m2, IV, q3weeks, Day 1 docetaxel 40mg/m2, IV, q3weeks, Day 1

SUMMARY:
Investigators assessed the effectiveness of HLX10, Trastuzumab and Chemotherapy in First-line Treatment of HER2-positive Recurrent/Metastatic Gastric Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven metastatic or locally advanced HER2-positive gastric cancer
2. Documented disease progression after receiving prior line of trastuzumab-containing chemotherapy for gastric cancer
3. Able and willing to give written informed consent and has signed the informed consent form (ICF), prior to performance of any trial activities.
4. Eligible male and female subjects aged ≥18 years.
5. Has measurable disease as determined by RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Has baseline left ventricular ejection fraction (LVEF) ≥ 55%.
8. Adequate organ function as demonstrated by laboratory test results within 14 days prior to first dose of study treatment.
9. Have urinary protein that is <2 on dipstick or routine urinalysis.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to first dose of study treatment.
11. Female subjects of childbearing potential and male subjects should be willing to use methods of birth control for the course of the study and up to 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Received prior anticancer treatment with targeted agents, chemotherapy, or radiotherapy within 14 days, with monoclonal antibodies within 28 days, has previously received treatment with ramucirumab, or has participated in another clinical trial within 14 days prior to start of study treatment.
2. Has experienced any Grade 3-4 gastrointestinal bleeding within 3 months prior to treatment.
3. Has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 3 months prior to treatment.
4. Has history of severe thromboembolism, including deep vein thrombosis and pulmonary embolism within 6 months prior to treatment.
5. Has an active or ongoing infection, symptomatic congestive heart failure, （6）uncontrolled angina pectoris, symptomatic or poorly controlled arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the investigator.

（7）Has ongoing or active psychiatric illness or social situation that would limit compliance with study requirements.

（8）Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

（9）Has evidence of active, non-infectious pneumonitis. （10）Have an elective or a planned major surgery during the course of the trial or has undergone major surgery within 4 weeks prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 18 months after start of treatment
  Progression-free survival in patients with HER2-positive gastric cancer receiving HLX10, trastuzumab, and chemotherapy combination treatment

SECONDARY OUTCOMES:
Overall survival | through study completion, an average of 2 years
  Overall survival
Objective response rate according to RECIST 1.1 | through study completion, an average of 2 years
  Objective response rate according to RECIST 1.1
Safety and tolerability based on incidence of treatment-emergent adverse events as assessed by CTCAE | Throughout the overall study period as well as up to 3 months after the last dose study treatment for each subject
  Safety and tolerability based on incidence of treatment-emergent adverse events as assessed by CTCAE